CLINICAL TRIAL: NCT03924024
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Orthopaedic Trauma Patients
Brief Title: rTMS for Orthopaedic Trauma Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: We never started the study due to logistical limitations.
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Nolan R, Assistant Professor, Director of Interventional Psychiatry Clinical Research, Department of Psychiatry and Behavioral Sciences, Stanford University Medical Center, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 49006
Record Dates: First submitted 2019-04-18; First posted 2019-04-23 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Orthopaedic Trauma
Keywords: Depression; Transcranial Magnetic Stimulation (TMS); Theta Burst; Orthopaedic Trauma; Pain
MeSH Terms: conditions — Depression; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Accelerated intermittent theta burst treatment (Experimental): All participants will receive accelerated intermittent theta-burst stimulation.
  Interventions: Device: Accelerated intermittent theta burst treatment

INTERVENTIONS:
Device: Accelerated intermittent theta burst treatment — All participants will receive accelerated intermittent theta-burst stimulation to the left DLPFC. Stimulation intensity will be standardized to 80% of resting motor threshold.
  Stimulation will be delivered to L-DLPFC using the Brainsway stimulator.

SUMMARY:
This study evaluates an accelerated schedule of theta-burst stimulation using a transcranial magnetic stimulation device for orthopaedic trauma patients. In this open label study, all participants will receive accelerated theta-burst stimulation. This study will examine whether symptoms of psychiatric distress and opioid use in orthopaedic trauma patients can be mitigated with rTMS to improve post-injury recovery.

DETAILED DESCRIPTION:
A large percentage of orthopaedic trauma patients suffer from psychiatric distress and chronic pain related to their injury and underlying psychosocial factors; this predicts poor post-injury recovery.

Repetitive transcranial magnetic stimulation (rTMS) is a neuromodulation technique used to stimulate areas of the brain that may modulate symptoms of pain, depression, and post-traumatic stress. The FDA-approved rTMS protocol for treatment is 10Hz stimulation for 40 minutes over the left dorsolateral prefrontal cortex (L-DLPFC) for the treatment of depression. This methodology has been very successful in real world situations, however poses some limitations, including the duration of the treatment session (approximately 40 minutes per treatment session). Recently, researchers have aggressively pursued modifying the treatment parameters to reduce treatment times with some preliminary success. This study will use modified parameters to create a more rapid form of treatment and look at outcome changes in pain and depression, commonly seen in orthopaedic trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 to 65 years of age.
* Able to provide informed consent.
* Present to Stanford Emergency Department as a trauma with a major operative lower extremity injury
* Glasgow coma scale of 15 within 24 hours after admission or extubation
* Negative urinary toxicology screen for illicit substances;
* Negative pregnancy test if female and less then 60 y/o;
* No suspicion for a head injury and/or negative head CT scan for intracranial hemorrhage or injury based on standard of care
* No history of seizure disorder or other neurological disorders.
* All patients included must screen positive for PHQ-9 score >4 (positive symptoms of depression) and CES-T score <36 (poor coping self-efficacy).

Exclusion Criteria:

* Incarceration,
* Pregnant females,
* Prior psychotic disorder,
* Current use of anti-depressant or anti-psychotic medications,
* Prior-admission opioid use within 30 days (patients will be screened for recent prescription opioid use using the CURES report),
* Heavy alcohol use,
* Lesional neurological disorder or brain implant or intracranial ferromagnetic material,
* Seizure disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the Hospital Anxiety and Depression Scale (HADS) | Baseline and immediate post-stimulation (up to 10 minutes to complete questionnaire)
  The Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) is a 14-item measure designed to assess anxiety and depression symptoms in medical patients, with emphasis on reducing the impact of physical illness on the total score. The depression items tend to focus on the anhedonic symptoms of depression. Items are rated on a 4-point severity scale (0 to 3). Overall scores range from 0 to 42, with lower scores corresponding to fewer symptoms. The HADS produces two scales, one for anxiety (HADS-A) and one for depression (HADS-D), differentiating the two states; each subscale score ranges from 0 to 21, with lower scores corresponding to fewer symptoms. Scores of greater than or equal to 11 on either HADS-A or HADS-D scales indicate a definitive case of anxiety and/or depression, respectively.

SECONDARY OUTCOMES:
Change from baseline in the Numeric Pain Rating Scale (NRS) | Baseline and immediate post-stimulation (up to 10 minutes to complete questionnaire)
  In a Numerical Rating Scale (NRS), patients are asked to make three pain ratings, corresponding to current, best and worst pain experienced over the past 24 hours.
  The average of the 3 ratings is used to represent the patient's level of pain over the previous 24 hours.
  Patients are asked to circle the number between 0 and 10 (first rating), 0 and 20 (second rating) and 0 and 100 (third rating) that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Change from baseline in the PTSD Checklist for DSM-5 (PCL-5) | Baseline and immediate post-stimulation (up to 10 minutes to complete questionnaire)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. It takes approximately 5-10 minutes to complete. It uses a 5-point Likert scale (0 = "Not at all" to 4 = "Extremely") to rate symptoms of PTSD. Scores can range from 0 to 60, with a cut-off score of 33 indicating a provisional diagnosis of PTSD until further psychometric work is available.
  The PCL-5 has a variety of purposes, including:
  1. Monitoring symptom change during and after treatment
  2. Screening individuals for PTSD
  3. Making a provisional PTSD diagnosis
  When necessary, the PCL-5 can be scored to provide a provisional PTSD diagnosis.
Change from baseline in the Trauma Coping Self-Efficacy (CSE-T) scale | Baseline and immediate post-stimulation (up to 10 minutes to complete questionnaire)
  9 item self-report scale designed to assess participants' capability of dealing with events following exposure to a traumatic event. Participants are asked to rate their ability from 1 "I'm not at all capable" to 7 "I'm totally capable". The lower the score, the more likely the participant is struggling to cope with their trauma.

CONTACTS AND LOCATIONS:
Overall Officials: Nolan Williams, MD, Principal Investigator — Stanford University
Locations (1):
- Department of Orthopaedic Surgery, Stanford Hospital, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data

REFERENCES:
- [Background] George MS, Lisanby SH, Avery D, McDonald WM, Durkalski V, Pavlicova M, Anderson B, Nahas Z, Bulow P, Zarkowski P, Holtzheimer PE 3rd, Schwartz T, Sackeim HA. Daily left prefrontal transcranial magnetic stimulation therapy for major depressive disorder: a sham-controlled randomized trial. Arch Gen Psychiatry. 2010 May;67(5):507-16. doi: 10.1001/archgenpsychiatry.2010.46. PMID 20439832
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Chung SW, Hill AT, Rogasch NC, Hoy KE, Fitzgerald PB. Use of theta-burst stimulation in changing excitability of motor cortex: A systematic review and meta-analysis. Neurosci Biobehav Rev. 2016 Apr;63:43-64. doi: 10.1016/j.neubiorev.2016.01.008. Epub 2016 Feb 3. PMID 26850210
- [Background] Jelic MB, Milanovic SD, Filipovic SR. Differential effects of facilitatory and inhibitory theta burst stimulation of the primary motor cortex on motor learning. Clin Neurophysiol. 2015 May;126(5):1016-23. doi: 10.1016/j.clinph.2014.09.003. Epub 2014 Sep 16. PMID 25281475
- [Background] Chung SW, Hoy KE, Fitzgerald PB. Theta-burst stimulation: a new form of TMS treatment for depression? Depress Anxiety. 2015 Mar;32(3):182-92. doi: 10.1002/da.22335. Epub 2014 Nov 28. PMID 25450537
- [Background] Plewnia C, Pasqualetti P, Grosse S, Schlipf S, Wasserka B, Zwissler B, Fallgatter A. Treatment of major depression with bilateral theta burst stimulation: a randomized controlled pilot trial. J Affect Disord. 2014 Mar;156:219-23. doi: 10.1016/j.jad.2013.12.025. Epub 2013 Dec 28. PMID 24411682
- [Background] Prasser J, Schecklmann M, Poeppl TB, Frank E, Kreuzer PM, Hajak G, Rupprecht R, Landgrebe M, Langguth B. Bilateral prefrontal rTMS and theta burst TMS as an add-on treatment for depression: a randomized placebo controlled trial. World J Biol Psychiatry. 2015 Jan;16(1):57-65. doi: 10.3109/15622975.2014.964768. Epub 2014 Nov 28. PMID 25430687
- [Background] Daskalakis ZJ. Theta-burst transcranial magnetic stimulation in depression: when less may be more. Brain. 2014 Jul;137(Pt 7):1860-2. doi: 10.1093/brain/awu123. Epub 2014 May 15. No abstract available. PMID 24833712
- [Background] Thut G, Pascual-Leone A. A review of combined TMS-EEG studies to characterize lasting effects of repetitive TMS and assess their usefulness in cognitive and clinical neuroscience. Brain Topogr. 2010 Jan;22(4):219-32. doi: 10.1007/s10548-009-0115-4. Epub 2009 Oct 28. PMID 19862614
- [Background] Holtzheimer PE 3rd, McDonald WM, Mufti M, Kelley ME, Quinn S, Corso G, Epstein CM. Accelerated repetitive transcranial magnetic stimulation for treatment-resistant depression. Depress Anxiety. 2010 Oct;27(10):960-3. doi: 10.1002/da.20731. PMID 20734360
- [Background] Fung PK, Robinson PA. Neural field theory of synaptic metaplasticity with applications to theta burst stimulation. J Theor Biol. 2014 Jan 7;340:164-76. doi: 10.1016/j.jtbi.2013.09.021. Epub 2013 Sep 21. PMID 24060620
- [Background] Greicius MD, Krasnow B, Reiss AL, Menon V. Functional connectivity in the resting brain: a network analysis of the default mode hypothesis. Proc Natl Acad Sci U S A. 2003 Jan 7;100(1):253-8. doi: 10.1073/pnas.0135058100. Epub 2002 Dec 27. PMID 12506194
- [Background] Greicius MD, Supekar K, Menon V, Dougherty RF. Resting-state functional connectivity reflects structural connectivity in the default mode network. Cereb Cortex. 2009 Jan;19(1):72-8. doi: 10.1093/cercor/bhn059. Epub 2008 Apr 9. PMID 18403396
- [Background] Hanlon CA, Dowdle LT, Austelle CW, DeVries W, Mithoefer O, Badran BW, George MS. What goes up, can come down: Novel brain stimulation paradigms may attenuate craving and craving-related neural circuitry in substance dependent individuals. Brain Res. 2015 Dec 2;1628(Pt A):199-209. doi: 10.1016/j.brainres.2015.02.053. Epub 2015 Mar 11. PMID 25770818
- [Background] Taylor JJ, Borckardt JJ, George MS. Endogenous opioids mediate left dorsolateral prefrontal cortex rTMS-induced analgesia. Pain. 2012 Jun;153(6):1219-1225. doi: 10.1016/j.pain.2012.02.030. Epub 2012 Mar 22. PMID 22444187
- [Background] Borckardt JJ, Weinstein M, Reeves ST, Kozel FA, Nahas Z, Smith AR, Byrne TK, Morgan K, George MS. Postoperative left prefrontal repetitive transcranial magnetic stimulation reduces patient-controlled analgesia use. Anesthesiology. 2006 Sep;105(3):557-62. doi: 10.1097/00000542-200609000-00020. PMID 16931989
- [Background] Borckardt JJ, Smith AR, Hutcheson K, Johnson K, Nahas Z, Anderson B, Schneider MB, Reeves ST, George MS. Reducing pain and unpleasantness during repetitive transcranial magnetic stimulation. J ECT. 2006 Dec;22(4):259-64. doi: 10.1097/01.yct.0000244248.40662.9a. PMID 17143157
- [Background] Borckardt JJ, Smith AR, Reeves ST, Weinstein M, Kozel FA, Nahas Z, Shelley N, Branham RK, Thomas KJ, George MS. Fifteen minutes of left prefrontal repetitive transcranial magnetic stimulation acutely increases thermal pain thresholds in healthy adults. Pain Res Manag. 2007 Winter;12(4):287-90. doi: 10.1155/2007/741897. PMID 18080048
- [Background] Borckardt JJ, Smith AR, Reeves ST, Madan A, Shelley N, Branham R, Nahas Z, George MS. A pilot study investigating the effects of fast left prefrontal rTMS on chronic neuropathic pain. Pain Med. 2009 Jul-Aug;10(5):840-9. doi: 10.1111/j.1526-4637.2009.00657.x. Epub 2009 Jul 6. PMID 19594842
- [Background] Borckardt JJ, Reeves ST, Weinstein M, Smith AR, Shelley N, Kozel FA, Nahas Z, Byrne KT, Morgan K, George MS. Significant analgesic effects of one session of postoperative left prefrontal cortex repetitive transcranial magnetic stimulation: a replication study. Brain Stimul. 2008 Apr;1(2):122-7. doi: 10.1016/j.brs.2008.04.002. PMID 19759838